CLINICAL TRIAL: NCT02330159
Title: A Feasibility Study of a Novel Technique for Pilonidal Wound Healing on Patient, Financial, and Quality of Life Outcomes
Brief Title: Feasibility of a Novel Technique for Pilonidal Wound Healing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast Clinical Research Associates, Houston, Texas (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: ACellCSA01
Record Dates: First submitted 2014-12-29; First posted 2015-01-01 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Pilonidal Disease; Pilonidal Cyst; Pilonidal Sinus
Keywords: Pilonidal; Quality of Life
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Novel Wound Healing Protocol: Subjects who have pilonidal disease that are being scheduled for surgical excision with our novel wound healing protocol. The disease can be actively infected or chronic.
  Interventions: Procedure: Novel Wound Healing Protocol

INTERVENTIONS:
Procedure: Novel Wound Healing Protocol — All patients will undergo surgical excision of the pilonidal disease and application of the novel wound healing protocol. After excision, MatriStem MicroMatrix powder will be applied to the wound bed. A MatriStem Multilayer Wound Matrix sheet will then be placed over the MatriStem MicroMatrix, secured in place, then covered with surface dressings. The wound should be left undisturbed for 10-14 days (until the 1st follow-up visit). At the 1st postoperative visit, the wound will reassessed, and a second application of the MicroMatrix to the wound bed may be performed. At subsequent follow-up visits at 1, 3, and 6 months, the wound bed will be measured, photo documentation will be captured, and patients will complete a survey to assess quality of life.

SUMMARY:
Pilonidal disease (PD) is a chronic disease with a major impact on patient quality of life and productivity. Thus, wound healing would have a significant effect on patient quality outcomes, patient quality of life, and healthcare utilization, as well as societal benefits from allowing this vital population to return to productivity. There is no consensus on postoperative wound care after surgery for PD. Negative pressure therapy is commonly used. However, this therapy is costly and cumbersome, and not evidence-based to optimize wound healing or postoperative patient or financial outcomes. The investigators goal is to investigate the impact of MatriStem® Wound Matrix and MicroMatrix® (ACell, Inc., Columbia, MD) on pilonidal wound healing. Secondary goals are to evaluate the impact of MatriStem Wound Matrix and MicroMatrix on postoperative outcomes, quality of life, and healthcare costs after surgical management of pilonidal disease.

DETAILED DESCRIPTION:
The investigators study has 2 main goals:

Aim 1: To evaluate wound healing at 2 weeks, 1 month, 3 months, and 6 months postoperatively in a prospective MatriStem Wound Matrix and MicroMatrix cohort

Aim 2: To evaluate pilonidal recurrence, reoperation rates, healthcare utilization, and quality of life at 2 weeks, 1 month, 3 months, and 6 months postoperatively in a prospective MatriStem Wound Matrix and MicroMatrix cohort

The investigators main hypothesis is that using MatriStem Wound Matrix and MicroMatrix for postoperative wound care will significantly improve healing rates, healthcare utilization, and quality of life outcomes. The null hypothesis of the study is that there is no significant difference in healing rates, healthcare utilization, and quality of life outcomes between MatriStem Wound Matrix/ MicroMatrix and negative pressure dressing cohorts. The alternative hypothesis is that there are differences in healing rates, healthcare utilization, and quality of life outcomes between MatriStem Wound Matrix/ MicroMatrix and negative pressure dressing cohorts.

Twenty consecutive patients undergoing surgical excision for Pilonidal Disease will be recruited for treatment. All patients will undergo comparable surgical excision and application of the novel protocol. The wound will be left undisturbed for 10-14 days (until the 1st follow-up visit). At the 1st scheduled postoperative visit, the wound will reassessed in the operative suite, and a second application of the protocol may be performed at the surgeon's discretion. The next follow-up visits will be at 1 month, 3 months, and 6 months. At these visits, the wound bed will be measured, photo documentation will be captured, and patients will complete a survey to assess quality of life.

Study Endpoints are:

1. Wound healing at 6 months. Success is defined at a 60% healing rate of epithelialization and wound contracture by volume measurements in centimeters.
2. Observation of quality of life, total costs for treatment, recurrence and reoperation rates at 6 months

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have pilonidal disease that are being scheduled for surgical excision
2. Subjects who are 18 years of age and older
3. Subjects of either gender
4. Subjects with no previous drainage or surgical procedures for pilonidal disease
5. Subjects who are willing and able to adhere to protocol requirements, agree to participate in the study program and provide written and informed consent.

Exclusion Criteria:

1. Subjects with previous drainage or surgical procedures for pilonidal disease.
2. Subjects who are pregnant.
3. Subjects with an allergy or medical condition that may interfere with the use of the study medications.
4. Subjects who have another condition or general disability or infirmity that in the opinion of the investigator precludes further participation in the study.
5. Patients under 16 years of age
6. Patients with incomplete medical records
7. Patients on chronic opioids for pain management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is patients with Pilonidal Disease undergoing surgical management. Patients will be recruited, evaluated in clinic preoperatively to assure they meet eligibility, then managed via a standard of care surgical procedure, with our protocol used for post-operative wound healing
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Wound Healing | 6 months
  To evaluate healing at 2 weeks, 1 month, 3 months, and 6 months postoperatively in a prospective MatriStem Wound Matrix and MicroMatrix cohort

SECONDARY OUTCOMES:
Healthcare costs using the novel protocol | 6 months
Quality of Life | 6 months
  To evaluate quality of life at 2 weeks, 1 month, 3 months, and 6 months postoperatively in a prospective MatriStem Wound Matrix and MicroMatrix cohort
Disease Recurrence | 6 months
  To evaluate recurrence and reoperation rates at 2 weeks, 1 month, 3 months, and 6 months postoperatively in a prospective MatriStem Wound Matrix and MicroMatrix cohort

CONTACTS AND LOCATIONS:
Overall Officials: Deborah S Keller, MS MD, Study Director — Colorectal Surgical Associates; Eric M Haas, MD, Principal Investigator — Colorectal Surgical Associates
Locations (1):
- Colorectal Surgical Associates, Houston, Texas, United States